CLINICAL TRIAL: NCT05206227
Title: Histamine as a Molecular Transducer of Adaptation to Exercise
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Uoregon_STUDY0000001; STUDY00000718 (CLOSED) (Other: University of Oregon); STUDY00000982 (CLOSED) (Other: University of Oregon); STUDY00001088 (CLOSED) (Other: University of Oregon)
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Postexercise Hypotension
Keywords: Histamine; Mast cell; Exercise
MeSH Terms: conditions — Post-Exercise Hypotension; Motor Activity | interventions — Exercise; Heating; Histamine Antagonists

STUDY DESIGN:
Intervention Model Description: This is a series of Basic Experimental Studies with Humans (BESH, as defined by PA-20-184). Subjects are enrolled (non-randomized) in different arms of the overall study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Aerobic Exercise (Experimental): Blood and skeletal muscle microdialysate collected during dynamic knee-extension exercise
  Interventions: Behavioral: Aerobic Exercise
- Heating (Experimental): Blood and skeletal muscle microdialysate collected during local and/or whole body heating
  Interventions: Drug: alpha-FMH
- Resistance and Aerobic Exercise (Experimental): Blood and urine collected during recovery from two modalities of exercise (This arm is now CLOSED)
  Interventions: Behavioral: Resistance and Aerobic Exercise
- Aerobic Exercise and Muscle Perfusion (Experimental): Muscle perfusion measured during aerobic exercise (This arm is now CLOSED)
  Interventions: Behavioral: Aerobic Exercise; Drug: Antihistamine

INTERVENTIONS:
Behavioral: Aerobic Exercise — Subjects will complete a single bout of aerobic exercise.
  Arms: Aerobic Exercise; Aerobic Exercise and Muscle Perfusion
Drug: alpha-FMH — Subjects will undergo either local heating with diathermy or whole body heating with far-infrared sauna.
  Other Names: Heating
  Arms: Heating
Behavioral: Resistance and Aerobic Exercise — Subjects will complete bouts of resistance and aerobic exercise.
  Arms: Resistance and Aerobic Exercise
Drug: Antihistamine — Subjects will complete a single bout of aerobic exercise under placebo vs antihistamine conditions.
  Arms: Aerobic Exercise and Muscle Perfusion

SUMMARY:
This study is investigating the role of histamine in generating adaptation to exercise

DETAILED DESCRIPTION:
Exercise promotes and maintains healthy cardiovascular, musculoskeletal, and metabolic function, but the signals and mechanisms which transduce these effects are poorly understood. Histamine plays a role in some of the positive benefits of exercise. The goal of this study is to determine the factors that regulate exercise's effects on endothelial and vascular function, with a focus on histamine released from mast cells in skeletal muscle. Participants will perform exercise or participate in interventions like heating that may replicate some of the effects of exercise. During most experiments, investigators will insert an intravenous catheter in an arm vein and microdialysis probes in the leg, collect dialysate from the microdialysis probe and blood from the vein, record noninvasive measures, and have the participants perform exercise or undergo heating.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -40

Exclusion Criteria:

* Systolic ≥ 120
* Diastolic ≥ 80
* Body mass index (BMI) ˃ 28 kg/m2
* Prior diagnosis of cardiovascular disease, diabetes, autonomic disorders, or asthma
* Smoking or nicotine use
* Ongoing medical therapy (other than birth control)
* Ongoing use of over-the-counter or prescription antihistamines
* Allergies or hypersensitivities to drugs, local anesthetics, skin disinfectants, adhesives, or latex
* Pregnant, breastfeeding subjects, or planning to become pregnant in the next 12 months
* Mobility restrictions that interfere with physical activity
* High physical activity based on International Physical Activity Questionaire (IPAQ1)
* Non-English speaking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of mast cell degranulation | One hour
  Beta-hexosaminidase release from mast cells in mast cell degranulation bioassay when exposed to intramuscular dialysate from exercising individuals
Histamine concentration | One hour
  Histamine concentration in intramuscular dialysate
Histamine metabolites | 24 hours
  Concentration of histamine metabolites in blood and urine
Muscle perfusion | One hour
  Skeletal muscle tissue oxygen index

CONTACTS AND LOCATIONS:
Overall Officials: John R Halliwill, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2026-01-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05206227/ICF_000.pdf